CLINICAL TRIAL: NCT01512199
Title: Randomized, Placebo Controlled, Double Blind Phase 1b/2 Study of U3-1287 (AMG 888) in Combination With Trastuzumab Plus Paclitaxel in Newly Diagnosed HER2 Positive Metastatic Breast Cancer (MBC)
Brief Title: Phase 1b/2 Study of U3-1287 in Combination With Trastuzumab Plus Paclitaxel in Newly Diagnosed Metastatic Breast Cancer (MBC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Improved, different standard of care caused business decision to terminate
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U31287-A-U202
Record Dates: First submitted 2012-01-09; First posted 2012-01-19 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Metastatic Breast Cancer
Keywords: U3-1287; Trastuzumab; Paclitaxel; newly diagnosed HER-2 positive; breast cancer; metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — patritumab; Trastuzumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- U3-1287 with trastuzumab + paclitaxel (Phase 1b) (Experimental): The Phase 1b portion is an open label, dose de escalation, single arm study designed to assess the safety and tolerability of up to 3 dose levels of U3- 1287 in combination with trastuzumab plus paclitaxel and will determine the recommended Phase 2 dose (RP2D) of U3 1287. The first cohort will receive U3- 1287 18 mg/kg intravenously (IV) in combination with trastuzumab plus paclitaxel once every 3 weeks (q3w).
  Interventions: Drug: U3-1287; Drug: Trastuzumab; Drug: Paclitaxel
- U3-1287 with trastuzumab+paclitaxel (Ph 2) (Experimental): The Phase 2 portion is a randomized, 2 arm, placebo controlled, double blind study designed to evaluate the safety and the efficacy of U3-1287 at the recommended phase 2 in combination with trastuzumab plus paclitaxel (experimental arm) relative to the control arm (trastuzumab plus paclitaxel and placebo).
  Interventions: Drug: U3-1287; Drug: Trastuzumab; Drug: Paclitaxel
- Placebo with trastuzumab+paclitaxel (Ph 2) (Placebo Comparator): The Phase 2 portion is a randomized, 2 arm, placebo controlled, double blind study designed to evaluate the safety and the efficacy of U3-1287 at the recommended phase 2 dose in combination with trastuzumab plus paclitaxel (experimental arm) relative to the control arm (trastuzumab plus paclitaxel and placebo).
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: U3-1287 — U3-1287: 18 mg/kg administered intravenously once every three weeks
  Arms: U3-1287 with trastuzumab + paclitaxel (Phase 1b)
Drug: Trastuzumab — Trastuzumab: 6 mg/kg up to 8 mg/kg administered intravenously once every three weeks
  Arms: U3-1287 with trastuzumab + paclitaxel (Phase 1b)
Drug: Paclitaxel — Paclitaxel: 175 mg/m^2 administered intravenously once every three weeks
  Arms: U3-1287 with trastuzumab + paclitaxel (Phase 1b)
Drug: U3-1287 — The maximum tolerated dose as determined in Phase 1b portion (between 9 mg/kg and 18 mg/kg) administered intravenously once every three weeks
  Arms: U3-1287 with trastuzumab+paclitaxel (Ph 2)
Drug: Trastuzumab — Trastuzumab: 6 mg/kg up to 8 mg/kg administered intravenously once every three weeks
  Arms: Placebo with trastuzumab+paclitaxel (Ph 2); U3-1287 with trastuzumab+paclitaxel (Ph 2)
Drug: Paclitaxel — Paclitaxel: 175 mg/m^2 administered intravenously once every three weeks
  Arms: Placebo with trastuzumab+paclitaxel (Ph 2); U3-1287 with trastuzumab+paclitaxel (Ph 2)
Drug: Placebo — Placebo: Dose corresponding to U3-1287 administered intravenously once every three weeks
  Arms: Placebo with trastuzumab+paclitaxel (Ph 2)

SUMMARY:
This is a Phase 1b/2 study. In Phase 1b portion, subjects will know the treatment they are receiving . Subjects will receive U3-1287 with trastuzumab plus paclitaxel . The phase 1b portion will determine if adding U3-1287 to trastuzumab plus paclitaxel will be safe in subjects with metastatic breast cancer. In phase 2 portion, subjects will be blinded to the treatments they are receiving . Subjects will receive either trastuzumab plus paclitaxel with U3-1287 or trastuzumab plus paclitaxel and placebo.The phase 2 portion will determine if adding U3-1287 to trastuzumab plus paclitaxel will be safe and improve survival in subjects with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy all of the following criteria to be included in the study:

1. Women ≥ 18 years old.
2. Histologically or cytologically confirmed adenocarcinoma of the breast with metastatic disease and at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) guidelines Version 1.1.
3. Documented HER2+ disease as measured by FISH or IHC (3+). See Appendix 17.8 for documentation criteria.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
5. Hematological function, as follows:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Platelet count >100 x 109/L
   * Hemoglobin ≥9 g/dL.
6. Renal function, as follows:

   - Calculated creatinine clearance ≥60 mL/min using the modified Cockcroft Gault equation.
7. Hepatic function, as follows:

   * AST ≤2.5 x ULN (if liver metastases are present, < 5 x ULN)
   * ALT ≤2.5 x ULN (if liver metastases are present, < 5 x ULN)
   * Alkaline phosphatase ≤ 2.0 x ULN (if bone or liver metastases are present, < 5 x ULN)
   * Bilirubin ≤1.5 x ULN.
8. Prothrombin time (PT) and partial thromboplastin time (PTT) ≤1.5 x ULN.
9. Availability of archived tumor sample or fresh tumor specimen (does not have to be provided by treatment start) to confirm HER2 status and for tumor biomarkers/mutation analysis.
10. Subjects must be postmenopausal (no menstrual period for a minimum of 12 months) or surgically sterile, or must use maximally effective birth control during the period of therapy, and be willing to use contraception for 6 months following the last investigational drug dose and have a negative urine or serum pregnancy test upon entry into this study if subject is of childbearing potential. Partners of subjects must be surgically sterile or willing to use a double barrier contraception method upon enrollment, during the course of the study, and for 6 months after last investigational drug dose received.
11. Subjects must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
12. Subjects must be competent and able to comprehend, sign, and date an IEC- or IRB-approved ICF before performance of any study specific procedures or tests.

Exclusion Criteria:

Subjects who meet any of the following criteria will be disqualified from entering the study:

1. Prior treatment for metastatic disease other than radiation therapy. Neoadjuvant/adjuvant therapy with paclitaxel, and/or docetaxel, and/or trastuzumab is allowed if completed more than 12 months prior to relapse/progression.
2. Clinically active brain metastases, defined as untreated symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Subjects with treated brain metastases that are no longer symptomatic and require no treatment with steroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy.
3. LVEF < 50%. History of LVEF decline to < 50% on prior trastuzumab therapy.
4. Therapeutic or palliative radiation therapy or major surgery within 4 weeks before study drug treatment.
5. History of other malignancies, except adequately treated nonmelanoma skin cancer, curatively treated in situ cancer, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years.
6. Uncontrolled hypertension (diastolic blood pressure > 100 mmHg or systolic blood pressure > 140 mmHg). Use of antihypertensive medications is permissible to maintain blood pressure within the required parameters.
7. Clinically significant electrocardiogram (ECG) changes that obscure the ability to assess the RR, PR, QT, QTc and QRS intervals.
8. Subjects with left bundle branch block, atrial fibrillation and use of a cardiac pacemaker specifically will be excluded.
9. Ascites or pleural effusion requiring chronic medical intervention.
10. Pre-existing peripheral neuropathy > grade 1.
11. Myocardial infarction, symptomatic CHF (New York Heart Association > Class II), unstable angina, or unstable cardiac arrhythmia requiring medication within 1 year before enrollment.
12. Use of cytochrome P450 (CYP) 3A4 (CYP3A4) or CYP2C8 inducers within 28 days prior to Day 1, use of CYP3A4 or CYP2C8 inhibitors within 14 days prior to Day 1, or concurrent use of CYP3A4 or CYP2C8 inducers or inhibitors (see Appendix 17.6 for list of CYP34A and CYP2C8 inhibitors and inducers).
13. Use of amiodarone within 6 months prior to enrollment.
14. Concurrent use of antiarrhythmic medications.
15. Participated in clinical drug studies within 4 weeks (2 weeks for small molecule tyrosine kinase inhibitors; 6 weeks for mitomycin C and nitrosoureas) before study drug treatment. Current participation in other investigational protocols or procedures.
16. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
17. Known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection.
18. History of hypersensitivity to any of the study drugs or to any excipients.
19. Serious intercurrent medical or psychiatric illnesses or any other conditions that in the opinion of the Investigator would impair the ability to give informed consent or unacceptably reduce protocol compliance or safety of the study treatment.
20. Pregnant, breastfeeding, or unwilling/unable to use acceptable contraception.
21. QTc interval > 450 msec by Friderica's formula on two successive screening measurements (second measurement is required if first measurement is > 450 msec.
22. Personal or family history of long-QT syndrome.
23. Subjects who are receiving drugs that may affect QTc (eg, quinidine or moxifloxacin).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2015-01-28 (Actual); Study Completion 2015-01-28 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose based on the incidence of dose limiting toxicities (phase 1b only) | Study start to approximately 16 weeks
  The following criteria will also be considered a dose limiting toxicity (DLT).
  * > 15% decrease in left ventricular ejection fraction (LVEF) from baseline or an LVEF value > 10% below lower limit of normal (LLN)
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 x the upper limit of normal (ULN) AND total bilirubin > 2 x ULN or international normalized ratio (INR) > 1.5
Progression Free Survival (Phase 2 only) | 52 weeks (Start to end of Phase 2)
  Tumor assessment will be conducted every 6 weeks independent of treatment cycle in accordance with Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)

SECONDARY OUTCOMES:
Pharmacokinetics (Area Under Curve) of U3-1287 when combined with trastuzumab plus paclitaxel | Pharmacokinetic blood samples will be taken on days 1, 2, 3, 8, 15, end of study (phase 1b) and during cycles 1-5, 9, 13, and at the end of study (Phase 2)
Pharmacokinetics (Area Under Curve Extrapolation Percent) of U3-1287 when combined with trastuzumab plus paclitaxel | Pharmacokinetic blood samples will be taken on days 1, 2, 3, 8, 15, end of study (phase 1b) and during cycles 1-5, 9, 13, and at the end of study (Phase 2)
Pharmacokinetics (C-max, C-min) of U3-1287 when combined with trastuzumab plus paclitaxel | Pharmacokinetic blood samples will be taken on days 1, 2, 3, 8, 15, end of study (phase 1b) and during cycles 1-5, 9, 13, and at the end of study (Phase 2)
Pharmacokinetics (T-max) of U3-1287 when combined with trastuzumab plus paclitaxel | Pharmacokinetic blood samples will be taken on days 1, 2, 3, 8, 15, end of study (phase 1b) and during cycles 1-5, 9, 13, and at the end of study (Phase 2)
Pharmacokinetics (Terminal Elimination Rate Constant) of U3-1287 when combined with trastuzumab plus paclitaxel | Pharmacokinetic blood samples will be taken on days 1, 2, 3, 8, 15, end of study (phase 1b) and during cycles 1-5, 9, 13, and at the end of study (Phase 2)
Pharmacokinetics (Terminal Half-Life) of U3-1287 when combined with trastuzumab plus paclitaxel | Pharmacokinetic blood samples will be taken on days 1, 2, 3, 8, 15, end of study (phase 1b) and during cycles 1-5, 9, 13, and at the end of study (Phase 2)
Pharmacokinetics (Volume of Distribution) of U3-1287 when combined with trastuzumab plus paclitaxel | Pharmacokinetic blood samples will be taken on days 1, 2, 3, 8, 15, end of study (phase 1b) and during cycles 1-5, 9, 13, and at the end of study (Phase 2)
Pharmacokinetics (Total Body Clearance) of U3-1287 when combined with trastuzumab plus paclitaxel | Pharmacokinetic blood samples will be taken on days 1, 2, 3, 8, 15, end of study (phase 1b) and during cycles 1-5, 9, 13, and at the end of study (Phase 2)
The best overall tumor response rate (Phase 1b) | Study start to 16 weeks
  The best overall tumor response is defined as the best response among all overall responses (in the order of Complete Response, Partial Response, Stable Disease, and Progressive Disease as per RECIST Version 1.1) recorded from the start of treatment.
Human anti-human antibody (HAHA) profile for U3-1287 (Phase 1b only) | Study start to 16 weeks
  The presence of HAHA (anti-U3-1287 neutralizing antibody) in serum will be assessed. To determine the presence of HAHA, blood samples will be taken preinfusion on Day 1 and at end of study treatment visit.
Human anti-human antibody (HAHA) profile for U3-1287 (Phase 2) | Study start to 52 weeks
  The presence of HAHA (anti-U3-1287 neutralizing antibody) in serum will be assessed. To determine the presence of HAHA, blood samples will be taken preinfusion on Day 1 of Cycles 1, 2, 3, 5, 9, and 13, and at end of study treatment visit.
Overall survival (Phase 2) | Study start to 52 weeks
Duration of response (Phase 2) | Study start to 52 weeks
Time to response (Phase 2) | Study start to 52 weeks
Time to progression (Phase 2) | Study start to 52 weeks
Duration of stable disease (Phase 2) | Study start to 52 weeks
The best overall tumor response rate (Phase 2) | Study start to 52 weeks
  The best overall tumor response is defined as the best response among all overall responses (in the order of Complete Response, Partial Response, Stable Disease, and Progressive Disease as per RECIST Version 1.1) recorded from the start of treatment.
Disease control rate (Phase 2) | Study start to 52 weeks
  The disease control rate is defined as the proportion of subjects with the best overall response of stable disease or better

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (8):
- Argentina (6):
  - Unidad de Investigación FP Clinical Pharma en Centro Medico Integral Fitz Roy, Acevedo, Buenos Aires F.D.
  - Centro Medico San Roque, San Miguel, Tucumán Province
  - Hospital Britanico, Buenos Aires
  - Sanatorio de la Providencia, Buenos Aires
  - Instituto Damic - Fundacion Rusculleda, Córdoba
  - ISIS Centro Especializado, Santa Fe
- Chile (2):
  - Instituto de Tereplas Oncologicas Providencia INTOP, Providencia, Santiago Metropolitan
  - Hospital Clinico San Borja Arriaran, Santiago